CLINICAL TRIAL: NCT04285515
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Assess the Efficacy and Safety of Lumateperone Monotherapy in the Treatment of Patients With Major Depressive Episodes Associated With Bipolar I or Bipolar II Disorder (Bipolar Depression) or Major Depressive Disorder
Brief Title: Clinical Trial Evaluating Lumateperone Monotherapy in the Treatment of Bipolar Depression or Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITI-007-403
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Bipolar Depression; Major Depressive Disorder
Keywords: Mixed Features
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major | interventions — lumateperone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lumateperone 42mg (Experimental): Lumateperone 42mg administered once daily in the evening
  Interventions: Drug: Lumateperone
- Placebo (Placebo Comparator): Matching placebo administered once daily in the evening
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Lumateperone — Lumateperone 42mg oral capsule
  Arms: Lumateperone 42mg
Drug: Placebos — Placebo oral capsule
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter study to evaluate the efficacy and safety of lumateperone monotherapy in the treatment of patients with major depressive episodes associated with Bipolar I or Bipolar II Disorder (Bipolar Depression) or major depressive disorder (MDD) who also meet the Diagnostic and Statistical Manual of Mental Disorder, 5th Edition (DSM-5) criteria for mixed-features. The study consists of a Screening Period, a Double-blind Treatment Period, and a Safety Follow-up Period.

ELIGIBILITY:
Major Inclusion Criteria:

* Male or female subjects of any race, ages 18-75 inclusive
* Meets the Diagnostic and Statistical Manual of Mental Disorder, 5th Edition (DSM 5) criteria for Bipolar I or Bipolar II Disorder or MDD
* The start of the current major depressive episode is at least 2 weeks but no more than 6 months prior to the Screening (Visit 1)
* Has at least moderate severity of illness, as measured by a rater-administered MADRS total score ≥ 24 and corresponding to a CGI S score of ≥ 4 at Screening (Visit 1) and Baseline (Visit 2)
* The patient meets the DSM-5 criteria for mixed-features specific to the Bipolar I or II diagnosis or MDD diagnosis
* Current major depressive episode is causing clinically significant distress or impairment in social, occupational, or other important areas of functioning
* Able to provide written informed consent

Major Exclusion Criteria:

* Any female subject who is pregnant or breast-feeding
* Any subject judged to be medically inappropriate for study participation
* The patient has a significant risk for suicidal behavior
* The patient presents with a lifetime history of epilepsy, seizure or convulsion, or electroencephalogram with clinically significant abnormalities, delirium, dementia, amnestic, or other cognitive disorder or significant brain trauma

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Kozauer, MD, Study Director — Intra-Cellular Therapies, Inc.
Locations (35):
- United States (13):
  - Clinical Site, Garden Grove, California
  - Clinical Site, Oceanside, California
  - Clinical Site, Sherman Oaks, California
  - Clinical Site, Lauderhill, Florida
  - Clinical Site, Miami, Florida
  - Clinical Site, Orange City, Florida
  - Clinical Site, Atlanta, Georgia
  - Clinical Site, Decatur, Georgia
  - Clinical Site, O'Fallon, Missouri
  - Clinical Site, Cedarhurst, New York
  - Clinical Site, New York, New York
  - Clinical Site, Charlotte, North Carolina
  - Clinical Site, Bellevue, Washington
- Bulgaria (8):
  - Clinical Site, Burgas
  - Clinical Site, Kardzhali
  - Clinical Site, Plovdiv
  - Clinical Site, Rousse
  - Clinical Site, Sofia
  - Clinical Site, Varna
  - Clinical Site, Veliko Tarnovo
  - Clinical Site, Vratsa
- Russia (4):
  - Clinical Site, Moscow
  - Clinical Site, Saint Petersburg
  - Clinical Site, Tomsk
  - Clinical Site, Yekaterinburg
- Serbia (3):
  - Clinical Site, Belgrade
  - Clinical Site, Kovin
  - Clinical Site, Kragujevac
- Ukraine (7):
  - Clinical Site, Kyiv
  - Clinical Site, Lviv
  - Clinical site, Odesa
  - Clinical Site, Odesa
  - Clinical Site, Poltava
  - Clinical Site, Smila
  - Clinical Site, Vinnytsia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Durgam S, Kozauer SG, Earley WR, Chen C, Huo J, Lakkis H, Stahl S, McIntyre RS. Lumateperone for the Treatment of Major Depressive Disorder With Mixed Features or Bipolar Depression With Mixed Features: A Randomized Placebo-Controlled Trial. J Clin Psychopharmacol. 2025 Mar-Apr 01;45(2):67-75. doi: 10.1097/JCP.0000000000001964. Epub 2025 Feb 14. PMID 39946099

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lumateperone 42mg | Placebo
Started | 243 | 245
Completed | 211 | 217
Not Completed | 32 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lumateperone 42mg | Placebo | Total
Number analyzed (Participants) | 240 | 241 | 481
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (14.54) | 43.4 (13.89) | 43.2 (14.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 148 | 298
  Male | 90 | 93 | 183
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 205 | 188 | 393
  Race: Black or African American | 32 | 49 | 81
  Race: Asian | 1 | 2 | 3
  Race: Other | 2 | 1 | 3
  Race: Multiple | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 82 | 78 | 160
  Ukraine | 20 | 17 | 37
  Bulgaria | 75 | 92 | 167
  Serbia | 15 | 24 | 39
  Russia | 48 | 30 | 78
Montgomery-Asberg Depression Rating Scale [Mean (Standard Deviation); unit: units on a scale] — Population: Numbers analyzed below represent all patients who received at least 1 dose of study drug and who had a nonmissing (predose) baseline assessment and at least 1 nonmissing postbaseline assessment of MADRS total score in the respective population.
  units on a scale
    Combined MDD and Bipolar Depression Mixed Features Population: number analyzed (Participants) | 192 | 191 | 383
    Combined MDD and Bipolar Depression Mixed Features Population | 31.3 (4.05) | 31.1 (4.07) | 31.3 (4.06)
    Bipolar Depression Mixed Features Population: number analyzed (Participants) | 100 | 99 | 199
    Bipolar Depression Mixed Features Population | 31.8 (4.40) | 31.1 (4.01) | 31.5 (4.22)
    MDD Mixed Features Population: number analyzed (Participants) | 92 | 92 | 184
    MDD Mixed Features Population | 30.8 (3.59) | 31.2 (4.16) | 31.0 (3.88)
    Overall Population: number analyzed (Participants) | 239 | 238 | 477
    Overall Population | 31.3 (4.33) | 31.4 (4.36) | 31.3 (4.34)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score
Description: The Montgomery-Åsberg Depression Rating Scale is a clinician-rated 10 item scale to assess depressive symptoms. Each item is rated on a 7-point scale from 0-6. The total score ranges from 0 to 60 with a higher score indicating increased severity of depressive symptoms.
Time Frame: Day 43
Population: Combined MDD and Bipolar Depression Mixed Features Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Lumateperone 42mg | Placebo
Number analyzed (Participants) | 192 | 191
score on a scale | -18.1 (0.71) | -12.4 (0.70)
Statistical Analysis 1: Comparison: Lumateperone 42mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Effects Model for Repeated Measure; Least Squares Mean Difference = -5.7, 95% CI 2-sided [-7.60 to -3.84], Standard Error of Mean 0.96

2. Primary Outcome: Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score
Description: as for outcome 1
Time Frame: Day 43
Population: Bipolar Depression Mixed Features Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Lumateperone 42mg | Placebo
Number analyzed (Participants) | 100 | 99
score on a scale | -17.7 (1.00) | -12.0 (0.96)
Statistical Analysis 1: Comparison: Lumateperone 42mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Effects Model for Repeated Measure; Least Squares Mean Difference = -5.7, 95% CI 2-sided [-8.29 to -3.05], Standard Error of Mean 1.33

3. Primary Outcome: Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score
Description: as for outcome 1
Time Frame: Day 43
Population: MDD Mixed Features Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Lumateperone 42mg | Placebo
Number analyzed (Participants) | 92 | 92
score on a scale | -18.2 (0.95) | -12.2 (0.96)
Statistical Analysis 1: Comparison: Lumateperone 42mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Effects Model for Repeated Measure; Least Squares Mean Difference = -5.9, 95% CI 2-sided [-8.61 to -3.29], Standard Error of Mean 1.35

4. Primary Outcome: Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score
Description: as for outcome 1
Time Frame: Day 43
Population: Overall Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Lumateperone 42mg | Placebo
Number analyzed (Participants) | 239 | 238
score on a scale | -17.7 (0.64) | -12.1 (0.63)
Statistical Analysis 1: Comparison: Lumateperone 42mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Effects Model for Repeated Measure; Least Squares Mean Difference = -5.6, 95% CI 2-sided [-7.25 to -3.88], Standard Error of Mean 0.86

5. Secondary Outcome: Clinical From Baseline in Clinical Global Impression Scale - Severity (CGI-S)
Description: The Clinical Global Impression Scale-Severity is a clinician-rated scale to assess a patient's overall mental health. The scale ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Day 43
Population: Combined MDD and Bipolar Depression Mixed Features Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Lumateperone 42mg | Placebo
Number analyzed (Participants) | 192 | 191
score on a scale | -1.8 (0.08) | -1.2 (0.08)
Statistical Analysis 1: Comparison: Lumateperone 42mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Effects Model of Repeated Measure; Least Squares Mean Difference = -0.6, 95% CI 2-sided [-0.81 to -0.39], Standard Error of Mean 0.11

6. Secondary Outcome: Clinical From Baseline in Clinical Global Impression Scale - Severity (CGI-S)
Description: as for outcome 5
Time Frame: Day 43
Population: Bipolar Depression Mixed Features Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Lumateperone 42mg | Placebo
Number analyzed (Participants) | 100 | 99
score on a scale | -1.8 (0.11) | -1.2 (0.11)
Statistical Analysis 1: Comparison: Lumateperone 42mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Effects Model for Repeated Measure; Least Squares Mean Difference = -0.6, 95% CI 2-sided [-0.91 to -0.31], Standard Error of Mean 0.15

7. Secondary Outcome: Clinical From Baseline in Clinical Global Impression Scale - Severity (CGI-S)
Description: as for outcome 5
Time Frame: Day 43
Population: MDD Mixed Features Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Lumateperone 42mg | Placebo
Number analyzed (Participants) | 92 | 92
score on a scale | -1.7 (0.11) | -1.1 (0.11)
Statistical Analysis 1: Comparison: Lumateperone 42mg vs Placebo; Test type: Superiority; p = 0.0003, Mixed Effects Model for Repeated Measure; Least Squares Mean Difference = -0.6, 95% CI 2-sided [-0.89 to -0.27], Standard Error of Mean 0.16

8. Secondary Outcome: Clinical From Baseline in Clinical Global Impression Scale - Severity (CGI-S)
Description: as for outcome 5
Time Frame: Day 43
Population: Overall Population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Lumateperone 42mg | Placebo
Number analyzed (Participants) | 239 | 238
score on a scale | -1.7 (0.07) | -1.1 (0.07)
Statistical Analysis 1: Comparison: Lumateperone 42mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Effects Model for Repeated Measure; Least Squares Mean Difference = -0.6, 95% CI 2-sided [-0.82 to -0.44], Standard Error of Mean 0.10

ADVERSE EVENTS:
Time Frame: From signing ICF until end of study procedures (~10 weeks), including 6 weeks of double-blind treatment.
Arm/Group | Lumateperone 42mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/240 | 0/241
Serious Adverse Events (participants affected / at risk) | 0/240 | 1/241
Other Adverse Events (participants affected / at risk) | 84/240 | 37/241
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lumateperone 42mg (N=240) | Placebo (N=241)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lumateperone 42mg (N=240) | Placebo (N=241)
Headache (Nervous system disorders) | 37 (37) | 30 (30)
Somnolence (Nervous system disorders) | 31 (31) | 4 (4)
Dizziness (Nervous system disorders) | 28 (28) | 4 (4)
Nausea (Gastrointestinal disorders) | 19 (19) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-01-27): https://cdn.clinicaltrials.gov/large-docs/15/NCT04285515/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/15/NCT04285515/SAP_001.pdf